CLINICAL TRIAL: NCT04088383
Title: A Prospective, Randomized, Double Blind Investigation of Amnios™ RT for the Treatment of Plantar Fasciitis
Brief Title: Amnios™ RT Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rev0
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amnios™ RT (Other)
  Interventions: Other: Amnios™ RT
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: Amnios™ RT — Acellular human allograft
  Arms: Amnios™ RT
Other: Saline — Sterile saline
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate clinical outcomes of patients with plantar fasciitis following treatment with Amnios™ RT. Patients will be randomized to either Amnios™ RT or a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of unilateral plantar fasciitis for ≥ 1 month (30 days) and ≤ 18 months by the Investigator
* VAS Foot Pain score of at least 45mm (out of 100mm scale) at randomization
* Plantar fasciitis with conservative treatment for ≥ 1 month (30 days), including any of the following modalities:

  * RICE
  * Stretching exercises
  * NSAIDs
  * Orthotics
* Diagnostic radiograph within 6 months of enrollment showing view of calcaneus, without evidence of calcaneal fracture or structural abnormalities
* BMI ≤ 40 kg/m2
* Age ≥ 18 years and < 80 years
* Willing and able to comply with the follow-up requirements of the protocol
* Signed an Informed Consent Form specific to this research and agreed to release of medical information

Exclusion Criteria:

* Prior surgery or trauma resulting in severe, permanent damage to the affected foot
* Require bilateral plantar fasciitis treatment at time of enrollment (with exception of compensatory symptoms on the non-affected foot)
* Prior use of any lower limb injection therapy, including corticosteroids or PRP in either foot within the last 3 months
* Has Type I or Type II diabetes mellitus
* Systemic disorders associated with enthesopathy (disorder of entheses, i.e. bone attachments) such as Gout, reactive arthritis, rheumatoid arthritis, etc.
* The presence of diagnosed comorbidities that can be confused with or can exacerbate the condition (as assessed by radiograph) including:

  * Calcaneal stress fracture
  * Nerve entrapment syndrome (diagnosed as Baxter Nerve Syndrome)
  * Fat pad atrophy (relative to expectations for patient's age)
  * Acute traumatic rupture of the plantar fascia
  * Calcaneal tumor
  * Tarsal tunnel syndrome (diagnosed)
  * Significant bone deformity of the foot that may interfere with the study
  * Other malignant tumors in the foot or conditions that may affect study outcomes
* Affected site exhibits clinical signs and symptoms of infection of the foot in question
* Known allergy or known sensitivity to aminoglycosides
* Non-ambulatory
* History of more than 14 days of treatment with immuno-suppressants (including systemic corticosteroids) or cytotoxic chemotherapy within 30 days prior to enrollment, or who are anticipated to require such medications during the course of the study
* Prior radiation at the site, with exception of diagnostic radiographs
* Use of any investigational drug(s) or investigational therapeutic device(s) within 3 months preceding enrollment
* Immune disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV)
* History of any condition (including drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol, in the judgment of the Investigator
* Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
* Prisoner

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Foot Pain Score | 3 Months
  The visual analog scale (VAS) is a patient questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "most intense pain imaginable" on the right border. The subject is instructed to place a vertical line on the scale that indicates the pain severity experienced; 0mm is equal to no pain and 100mm is most intense pain imaginable. Study staff records the distance of the patient's mark on the scale in millimeters.
Serious Adverse Events | 12 Months
  The occurrence of serious adverse events that are related to the product.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-X-Cell Research, San Antonio, Texas, United States